CLINICAL TRIAL: NCT06235281
Title: A Single-Arm, Open-Label, Pilot Study of Concurrent Phototherapy and POTELIGEO (Mogamulizumab-kpkc) in Early Stage Mycosis Fungoides (PLIGHT)
Brief Title: Phototherapy and Mogamulizumab in Early Stage MF (PLIGHT)
Acronym: PLIGHT
Status: Suspended | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Kyowa Hakko Kirin Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-21143
Record Dates: First submitted 2024-01-23; First posted 2024-01-31 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Mycosis Fungoides
Keywords: Early Stage Mycosis Fungoides
MeSH Terms: conditions — Mycosis Fungoides | interventions — mogamulizumab; Phototherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- POTELIGEO & Phototherapy combination therapy (Experimental): POTELIGEO (mogamulizumab-kpkc) will be given according to FDA approved dose and scheduled for 8 cycles. After 2 cycles of POTELIGEO, all subjects will start phototherapy as combination therapy.
  Interventions: Drug: Mogamulizumab-Kpkc; Device: Phototherapy

INTERVENTIONS:
Drug: Mogamulizumab-Kpkc — Participants will receive 8 total cycles of Mogamulizumab-Kpkc over approximately 224 days.
  Other Names: POTELIGEO
Device: Phototherapy — Participants will begin receiving Phototherapy on day 56 and will continue until day 224. Participants with Complete response (CR) or Partial response (PR) to therapy at day 224 will remain on phototherapy maintenance.
  Other Names: nb-UVB

SUMMARY:
This is an open label, single arm, single-center, pilot study of concurrent phototherapy and POTELIGEO (mogamulizumab-kpkc) in early-stage mycosis fungoides.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent/assent for the trial.
* Be at least 18 years of age on day of signing informed consent.
* Able to adhere to the study visit schedule and other protocol requirements.
* Diagnosis of mycosis fungoides (MF) based on a combination of histological, clinical, and immunophenotypical criteria. The histological criteria will be based on skin biopsy from the most representative skin area.
* CTCL (Mycosis fungoides) stage IA-IIA (early stage) at the time of screening with either B0 blood involvement with a positive T-cell receptor (TCR) gene rearrangement or B1 blood involvement with positive TCR gene rearrangement. The TNMB system will be used to classify the stage of disease.
* Any number of prior therapies is allowed.
* Patients must have stable disease (SD), partial response (PR) or disease progression (PD) after 3 or more months prior to date of consent of one of the following treatments: Phototherapy [narrow-band ultraviolet B (nb-UVB) or Psoralen ultraviolet A (PUVA)] alone or PUVA in combination with topical therapy such as nitrogen mustard, steroids, or bexarotene gel progression of skin disease on long-term maintenance phototherapy.
* A minimum washout period of 14 days prior after previous CTCL therapy before the first day of treatment.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Subjects on a stable dose of a low dose systemic corticosteroid (≤ 20 mg prednisone equivalent) for at least 4 weeks prior to day 1 of treatment may continue use. Investigator should attempt to taper the use to the lowest dosage tolerable while on study. Initiation of treatment with systemic corticosteroids or increase in dose while on study is not permitted except to treat an infusion reaction. Subjects may receive intra-articular corticosteroid injections, intraocular corticosteroid drops, inhalation or nasal corticosteroids and replacement doses of systemic corticosteroids as needed.
* Subjects on a stable dose of topical calcineurin inhibitors, medium or low potency topical corticosteroids for at least 4 weeks prior to the consent date may continue use at the same dose, although the investigator should attempt to taper the use to the lowest dosage tolerable while on study. Initiation of treatment with topical corticosteroids while on study is not permitted except to treat an acute rash.
* Resolution of all clinically significant toxic effects of prior cancer therapy to Grade ≤ 1 by the National Cancer Institute Common Terminology Criteria for Adverse Events, version 5.0 (NCI-CTCAE, v.5.0).
* Laboratory parameters required to be met prior to the initiation of each cycle: A) Adequate hepatic and kidney function defined as Serum bilirubin less than 1.5x upper limit of normal (ULN), AST and ALT must be less than 2.5x ULN, Serum creatinine < 1.5x upper limit of normal (ULN) OR calculated creatinine clearance ≥ 60 mL/min using the Cockcroft-Gault formula. B) Adequate hematological function defined as Serum Platelets greater than or equal to 100,000/mm3, Hemoglobin greater than or equal to 9g/dL without transfusion support and Absolute neutrophil count (ANC) greater than or equal to 1,500 cells/μL (greater than or equal to 1,500/mm3).
* Subjects previously treated with POTELIGEO (mogamulizumab-kpkc) are eligible if they achieved complete response on mogamulizumab and the last treatment was over 1 year ago.
* Female of childbearing potential (FCBP) must have a negative pregnancy test within 7 days of receiving study medication.
* Male subjects and their female partners of childbearing potential must be willing to use an appropriate method of contraception defined as oral contraceptives, double barrier method (condom plus spermicide or diaphragm plus spermicide) or practice true abstinence from sexual intercourse (periodic abstinence, e.g., calendar, ovulation, symptothermal, post-ovulation methods and withdrawal are not acceptable methods of contraception) during the study and for 3 months after the last dose.

Exclusion Criteria:

* Current evidence of large cell transformation (LCT) on biopsy. Subjects with clinical features suggestive of LCT must have a biopsy performed within 4 months prior to Cycle

  1 Day 1 to rule out transformed disease. Subjects with a history of LCT but without current aggressive disease and no current evidence of LCT on pathology in skin or lymph nodes would be eligible.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator (including but not limited to severe dermatitis). Any active infection requiring systemic therapy, including human immunodeficiency virus (HIV), human T-cell lymphotropic virus (HTLV), Hepatitis B, and/or Hepatitis C.
* Active herpes simplex or herpes zoster. Subjects on prophylaxis for herpes who started taking medication at least 30 days prior to consent, and have no active signs of active infection, and whose last active infection was more than 6 months ago, may enter the study, and should continue to take the prescribed prophylactic medication for the duration of the study.
* Any major surgery or radiation therapy within four weeks.
* Diagnosed with a malignancy in the past 2 years except nonmelanoma skin cancers, melanoma in situ, localized cancer of the prostate with current prostate-specific antigen of less than 0.1 ng/mL, treated thyroid cancer, cervical carcinoma in situ or ductal/lobular carcinoma in situ of the breast with in the past 2 years may enroll as long as there is no current evidence of active disease.
* If pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the trial, starting with consent through 30 after the last dose of trial treatment.
* Significant uncontrolled intercurrent illness including, but not limited to: uncontrolled infection requiring systemic antibiotics; clinically significant cardiac disease (class III or IV of the New York Heart Association [NYHA] classification); unstable angina pectoris; angioplasty, stenting, or myocardial infarction within 6 months; uncontrolled hypertension (systolic blood pressure (BP) greater than 160 mm Hg or diastolic BP greater than 100 mm Hg, found on 2 consecutive measurements separated by a 1-week period) despite 2 anti-hypertensive medications; clinically significant cardiac arrhythmia or uncontrolled diabetes.
* Known active autoimmune disease will be excluded. (For example, Graves' disease; systemic lupus erythematosus; rheumatoid arthritis; Crohn's disease).
* Documented prior hypersensitivity (i.e., allergic reaction) to POTELIGEO (mogamulizumab-kpkc) with a severity of Grade 2 or higher.
* Experienced allergic (does not include a grade 1-2 infusion-related) reactions to monoclonal antibodies or other therapeutic proteins.
* History of allogeneic transplant or autologous hematopoietic stem cell transplant.
* Subjects on any immunomodulatory drug for concomitant or intercurrent conditions other than T-cell lymphoma or who have received any of these agents within 4 weeks of treatment, including but not limited to the following, will be excluded: low dose or oral methotrexate; azathioprine; iv immunoglobulin; low dose or oral cyclophosphamide; cyclosporine; mycophenolate; infliximab; etanercept; leflunomide; adalimumab; lenalidomide; abatacept; rituximab; anakinra; interferon-β; IL-2 and natalizumab.
* Currently taking potential photosensitizing medications.
* Known or symptoms of photosensitivity disorders, including porphyria, lupus erythematosus, xeroderma pigmentosum, vitiligo, etc.
* History of phototoxic eruptions, photoallergic eruptions or PMLE (polymorphous light eruption).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-18 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | 225 days
  Overall Response Rate (ORR) is defined as the total proportion of patients in Complete Response (CR) + Partial Response (PR) and will be evaluated at days 57 and 225.

SECONDARY OUTCOMES:
Time to response in skin | 225 days
  Date of initiation of treatment to date when criteria for response (PR or CR) first met.
Duration of skin response for responding subjects | 5 years
  Date when criteria for response (CR or PR) first met until date response first lost; date of loss of response = date when first meets criteria for PD or relapse.
Time to treatment failure | 5 years
  Date of initiation of treatment until abandonment of therapy or the addition of another mycosis fungoides specific therapy.
CD4+CD26- and CD4+CD7 Change | 5 years
  This will be defined as the Change from baseline and longitudinally during the study in absolute numbers of CD4+CD26- and CD4+CD7- in PBC by 10 color flow cytometry.
Pruritus Change | 5 years
  This will be defined as the change from baseline and longitudinally during the study in Pruritus, by quantification of pruritus severity by a visual analog scale.

CONTACTS AND LOCATIONS:
Overall Officials: Lubomir Sokol, MD, PhD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States